CLINICAL TRIAL: NCT05527730
Title: Clinical Trial Evaluating Outcomes of Self-Fit and Professionally Fit Hearing Aids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Whisper.ai (Industry)
Collaborators: San Jose State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DM0224
Record Dates: First submitted 2022-07-21; First posted 2022-09-02 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hearing Loss
Keywords: Self-fitting hearing aids; conventional hearing aid fitting
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: This multi-center, prospective, randomized cross-over clinical trial compares two methods of fitting individuals with hearing loss with a therapeutic amplification device (i.e., hearing aids). Subjects will wear the Whisper Hearing System for the PRO-FIT and SELF-FIT for two weeks each, totalling to approximately 1 month of wear throughout the trial.
Who Masked: Participant
Masking Description: The participant were be blind folded for the type of fitting for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Screening, intake and first fit (either PRO-FIT or SELF-FIT fitting ) (Active Comparator): This multi-center, prospective, randomized cross-over clinical trial compares two methods of fitting individuals with hearing loss with a therapeutic amplification device (i.e., hearing aids). Subjects will wear the Whisper Hearing System for the PRO-FIT and SELF-FIT for two weeks each, totalling to approximately 1 month of wear throughout the trial. At the first visit, all individuals will go through intake procedures and a basic audiologic evaluation. After this is completed, individuals are randomized into one of two arms of the study Individuals in the first visit of the study will receive the conventional PRO-FIT method for the first two weeks, then will switch to the experimental SELF-FIT method for the last half of the study.
  Interventions: Device: Comparison of PRO-FIT or SELF-FIT fitting
- Second fit (either PRO-FIT or SELF-FIT fitting ) (Sham Comparator): Conversely, individuals in the second visit of the study will receive the experimental SELF-FIT method for the first two weeks, then will switch to the conventional PRO-FIT method for the last two weeks. The two fitting methods (PRO-FIT and SELF-FIT) will be compared to evaluate the efficiency and reliability of the Whisper hearing system self-fitting algorithm.
  Interventions: Device: Comparison of PRO-FIT or SELF-FIT fitting

INTERVENTIONS:
Device: Comparison of PRO-FIT or SELF-FIT fitting — add
  Other Names: SELF-FIT fitting; PRO-FIT fitting

SUMMARY:
Approximately 48 million people in the United States have hearing loss or hearing difficulties in noisy environments. Whisper.ai Inc has previously brought to market a commercial hearing aid system that reduces background noise and amplifies voices and sounds of interest using its proprietary platform based on machine learning and artificial intelligence technologies.

Whisper.ai Inc now seeks to bring to market a new hearing system that will incorporate a "self-fitting" capability. Self-fitting hearing aids have emerged in recent years as a potentially viable option to calibrate hearing aids to the needs of individual users without clinician intervention. The purpose of this project is to evaluate the efficiency and reliability of the fitting procedure and algorithms developed by Whisper.ai Inc. The study will be carried out using a randomized crossover design in two phases: in phase 1, subjects will be tested and a hearing aid will be fitted using conventional audiological standard procedures , and in phase 2, the subject will be tested and a hearing aid will be fitted using the results of the self-fitting algorithm.

Objective, subjective, and behavioral responses will be gathered from a variety of hearing-related surveys and tests, and will be analyzed quantitatively to evaluate the efficiency and reliability of the self-fitting algorithm. The investigators expect the fitting results of the Whisper.ai self-fitting algorithm to be similar to those of standardized fitting procedures conducted by hearing professionals.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-80 years old
* Mild-to-moderate hearing loss in both ears from 500 to 4000 Hz
* Reported one year of previous hearing aid experience in at least one ear
* Ability to use a laptop/desktop computer to browse the internet
* Ability to complete online surveys in a web browser
* Communicates verbally and in writing in English

Exclusion Criteria:

* History of neurological deficits (e.g. stroke, Alzheimer's disease, etc.)
* Inability to remain alert throughout initial testing appointment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Hearing aid gain comparisons using Real Ear Measures Data Analysis Plan | 4 weeks
  To evaluate, fine-tune, and compare the gains produced by the Whisper Hearing System using both PRO-FIT and SELF-FIT, general standard-of-care real-ear measurements (REM) will be used. Real Ear Measures (REMs) provide an objective measure of sound pressure level in an individual's ear canal. Frequencies critical to speech understanding (500 through 4000 Hz) will be averaged to yield a single value similar to a pure tone average. A mean absolute difference will be used to evaluate whether the SELF-FIT is non-inferior to the PRO-FIT; a mean absolute difference less than 5 dB will be considered as a non-significant difference when comparing REMs between the SELF-FIT and PRO-FIT groups.

SECONDARY OUTCOMES:
Speech perception scores comparison | 2 hours for the testing, 4 weeks trial
  The Quick Speech In Noise (QuickSIN) will provide a behavioral measure that will be compared across fitting conditions.The outcome of a non-inferiority trial may be assessed by a two-sided t-test, using a 95% confidence interval. A two-sided t-test will be used to compare the two final Quick Speech in Noise scores across fitting groups.Minimum value: -4.5 SNR Loss Maximum value: 25.5 SNR Loss Lower score here is better performance/outcome (-4.5 is the best possible score).
Overall perception hearing | 4 weeks
  Abbreviated Profile of Hearing Aid Benefit (APHAB) is a 24-item self-assessment inventory in which subjects report the amount of trouble they are having with communication or noises in various everyday situations. The APHAB produces scores for 4 subscales: Ease of Communication, Reverberation, Background Noise, and Aversiveness. These are combined to create a global score, which will be used to evaluate the overall benefit of amplification for each fitting strategy (SELF-FIT and PRO-FIT).
  The outcome of a non-inferiority trial may be assessed by a two-sided t-test, using a 95% confidence interval. A two-sided t-test with 95% confidence intervals will be used to determine whether APHAB outcomes differ between the SELF-FIT and the PRO-FIT.
  Minimum value: 0% of problems Maximum value: 100% of problems Lower score here is a lower percent of problems, or better performance/outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Whisper.ai, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No